CLINICAL TRIAL: NCT04194541
Title: Wound Dressings for Hidradenitis Suppurativa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hadar Lev-Tov, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20191046
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Group (Experimental): Participants will be provided a kit containing 3 dressings: Cutimed Sorbact Hydroactive B, Cutimed Siltec, and Sorbion Sana multi-star. Participant can use their dressing of choice and can change their dressings as needed for 6 consecutive weeks.
  Interventions: Device: Cutimed Sorbact Hydroactive B wound dressing; Device: Cutimed Siltect wound dressing; Device: Sorbion Sana multi-star wound dressing

INTERVENTIONS:
Device: Cutimed Sorbact Hydroactive B wound dressing — Wound dressing applied and changed as needed.
Device: Cutimed Siltect wound dressing — Wound dressing applied and changed as needed.
Device: Sorbion Sana multi-star wound dressing — Wound dressing applied and changed as needed.

SUMMARY:
The primary purpose of this research is to determine how the types of wound dressings affect quality of life for people with Hidradenitis Suppurativa (HS).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age
* Diagnosed with Hidradenitis Suppurativa (all stages of disease) by Dermatologist
* Presence of at least one lesion with active drainage
* Willing and able to provide informed consent

Exclusion Criteria:

* Subjects younger than 18-years-old.
* Prisoners
* Pregnant or lactating women
* Adults unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Lev-Tov, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were assigned to receive all three wound dressings and can choose to use whichever dressing they prefer. Each participant can have one or multiple wounds/lesions. Whether each participant had one or multiple of wounds/lesions was not data of interest. This information was not collected and included in the data analysis.
Period: Visit 0 (Baseline)
Arm/Group | Treatment Group
Started | 28
Completed | 28
Not Completed | 0
Period: Day 1 Through 13
Arm/Group | Treatment Group
Started | 28
Completed | 19
Not Completed | 9
Not completed — Lost to Follow-up | 3
Not completed — Coronavirus Disease of 2019 (COVID-19) shut down | 6
Period: Visit 1 (Day 14)
Arm/Group | Treatment Group
Started | 19
Completed | 19
Not Completed | 0
Period: Day 15 Through Week 6
Arm/Group | Treatment Group
Started | 19
Completed | 14
Not Completed | 5
Not completed — Lost to Follow-up | 5
Period: Visit 2 (6 Weeks)
Arm/Group | Treatment Group
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.57 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Dermatology Life Quality Index (DLQI) Scores
Description: Participant quality of life as measured via DLQI. DLQI has a total score ranging from 0-30 with the higher score indicating more impairment on the participant's quality of life.
Time Frame: At Baseline, at 6 Weeks
Population: Data is representative of the 14 participants that completed the study per protocol (completed Week 6 visit).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
score on a scale
  Visit 0 (Baseline) | 15.5 [11 to 24]
  Visit 2 (Week 6) | 12.5 [7.8 to 15]

2. Secondary Outcome: Average Pain as Assessed by the Numerical Rating Scale (NRS)
Description: The average pain reported over the last 24 hours will be measured using the NRS with scores ranging from 0-10 with the higher score indicating more severe pain.
Time Frame: At Baseline, at 6 Weeks
Population: Data is representative of the 14 participants that completed the study per protocol (completed Week 6 visit).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
score on a scale
  Visit 0 (Baseline) | 6.5 [3 to 7.5]
  Visit 2 (week 6) | 5 [2.75 to 7.25]

3. Secondary Outcome: Maximal Pain as Assessed by the Numerical Rating Scale (NRS)
Description: The pain rating at its worse over the last 24 hours will be reported as the maximal pain using the NRS with scores ranging from 0-10 with the higher score indicating more severe pain.
Time Frame: At Baseline, at 6 Weeks
Population: Data is representative of the 14 participants that completed the study per protocol (completed Week 6 visit).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
score on a scale
  Visit 0 (Baseline) | 7.5 [3.5 to 8]
  Visit 2 (Week 6) | 6.5 [2.75 to 7.25]

4. Secondary Outcome: Sleep Rating
Description: Sleep rating will be evaluated using a 5 point Likert scale ranging from 1-5 with the higher score indicating increased sleep disturbance.
Time Frame: At Baseline, at 6 Weeks
Population: Data is representative of the 14 participants that completed the study per protocol (completed Week 6 visit).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
score on a scale
  Visit 0 (Baseline) | 4 [2 to 4]
  Visit 2 (Week 6) | 3.5 [1.75 to 3.5]

5. Secondary Outcome: Drainage Rating
Description: Lesion drainage rating will be evaluated using a 4 point Likert scale ranging from 1-4 with the higher score indicating increased lesion draining. For participants with multiple wounds/lesions, the drainage rating will be a comprehensive assessment of all wounds/lesions.
Time Frame: At Baseline, at 6 Weeks
Population: Data is representative of the 14 participants that completed the study per protocol (completed Week 6 visit).
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
score on a scale
  Visit 0 (Baseline) | 3.06 [3 to 4]
  Visit 2 (Week 6) | 3.6 [3 to 4]

6. Secondary Outcome: Odor Rating
Description: Lesion odor rating will be evaluated using a 4 point Likert scale ranging from 1-4 with the higher score indicating increased lesion odor. For participants with multiple wounds/lesions, the odor rating will be a comprehensive assessment of all wounds/lesions.
Time Frame: At Baseline, at 6 Weeks
Population: Data is representative of the 14 participants that completed the study per protocol (completed Week 6 visit).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
score on a scale
  Visit 0 (Baseline) | 2.5 [2 to 3]
  Visit 2 (Week 6) | 2.5 [2 to 3.5]

7. Secondary Outcome: Number of Participants at Each Hidradenitis Suppurativa Physician Global Assessment (HS-PGA) Grading
Description: HS-PGA Scale scores patient disease severity as one of the following: clear, minimal, mild, moderate, severe, and very severe. The number of participants scored at each scale will be reported.
Time Frame: At 6 Weeks
Population: Data is representative of the 14 participants that completed the study per protocol (completed Week 6 visit).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
Participants
  Clear | 0
  Minimal | 0
  Mild | 0
  Moderate | 10
  Severe | 3
  Very Severe | 1

8. Secondary Outcome: Average Frequency of Dressing Changes
Description: Participant reported frequency of dressing changes per wound per day. For participants with multiple wounds/lesions, the frequency of dressing changes will be a comprehensive assessment of all wounds/lesions.
Time Frame: 6 Weeks
Population: Only 1 participant returned their survey for this outcome
Measure: Mean (Inter-Quartile Range); unit: dressing changes per wound per day
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
dressing changes per wound per day | 1 [1 to 1]

9. Secondary Outcome: Number of Participants Reporting Overall Dressing Preference for Specific Body Part
Description: Overall dressing preference will be reported as the number of participants preferring to use a particular wound dressing in the kit provided.
Time Frame: At Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 28
Participants
  Cutimed Sorbact Hydroactive B Wound Dressing | 9
  Cutimed Siltect Wound Dressing | 13
  Sorbion Sana Multi-star Wound Dressing | 6

10. Secondary Outcome: Number of Participants Reporting Dressing Preference for Each Specific Body Part
Description: Participant reported dressing preference for specific body parts for each of the interventions received.
Time Frame: Visit 1 (Day 14)
Population: Not all participants have wounds in all body parts noted (axilla, buttocks, groin, abdomen and breast).
Measure: Count of Participants; unit: Participants
Groups:
- Cutimed Sorbact Hydroactive B; Cutimed Siltect; Sorbion Sana Multi-Star: All participants received all three interventions (Cutimed Sorbact Hydroactive B, Cutimed Siltect and Sorbion Sana Multi-Star)
Arm/Group | Cutimed Sorbact Hydroactive B | Cutimed Siltect | Sorbion Sana Multi-Star
Number analyzed (Participants) | 19 | 19 | 19
Participants
  Axilla | 7 | 8 | 4
  Buttocks/gluteal fold | 1 | 3 | 2
  Groin | 2 | 1 | 1
  Abdomen | 1 | 2 | 0
  Breast/inframammary fold | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks.
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT04194541/Prot_SAP_000.pdf